CLINICAL TRIAL: NCT01648582
Title: The Efficacy and Safety of Once-Weekly, Subcutaneous Dulaglutide Compared to Once-Daily Insulin Glargine in Patients With Type 2 Diabetes Mellitus on Metformin and/or a Sulfonylurea
Brief Title: A Study Comparing the Effects and Safety of Dulaglutide With Insulin Glargine in Type 2 Diabetes Mellitus
Acronym: AWARD-CHN2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13439; H9X-CR-GBDK (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-16; First posted 2012-07-24 (Estimated); Results first posted 2015-07-24 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dulaglutide; Insulin Glargine; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1.5 mg Dulaglutide (Experimental): 1.5 milligrams (mg) dulaglutide administered as one subcutaneous (SC) injection once-weekly added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea for up to 52 weeks. Participants are blinded to the dulaglutide dose.
  Interventions: Drug: Dulaglutide; Drug: Metformin; Drug: Sulfonylureas
- 0.75 mg Dulaglutide (Experimental): 0.75 mg Dulaglutide administered as one SC injection once-weekly added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea for up to 52 weeks. Participants are blinded to the dulaglutide dose.
  Interventions: Drug: Dulaglutide; Drug: Metformin; Drug: Sulfonylureas
- Insulin Glargine (Active Comparator): Insulin glargine administered based on fasting blood glucose concentrations per the dosing titration schedule as once daily SC injection at bedtime added to participant's pre-study prescribed dose of metformin and /or a sulfonylurea for up to 52 weeks.
  Interventions: Drug: Insulin glargine; Drug: Metformin; Drug: Sulfonylureas

INTERVENTIONS:
Drug: Dulaglutide — Administered SC
  Other Names: LY2189265
  Arms: 0.75 mg Dulaglutide; 1.5 mg Dulaglutide
Drug: Insulin glargine — Administered SC per dosing titration schedule
  Arms: Insulin Glargine
Drug: Metformin — Administered orally at pre-study prescribed dose, and is not being provided as part of the trial.
Drug: Sulfonylureas — Administered orally at pre-study prescribed dose, and is not being provided as part of the trial.

SUMMARY:
The purpose of this study is to examine if once-weekly dulaglutide is efficient and safe compared to once-daily insulin glargine in participants with type 2 diabetes mellitus who have inadequate glycemic control with 1 or 2 oral antihyperglycemic medications (OAM) (metformin and/or a sulfonylurea), in addition to any healthy lifestyle changes recommended by their healthcare providers.

ELIGIBILITY:
Inclusion Criteria:

* Have type 2 diabetes mellitus for at least 6 months
* Have been taking metformin and/or a sulfonylurea for at least 3 months before screening and have been on a stable therapeutic dose for at least 8 weeks
* Glycosylated hemoglobin (HbA1c) value of ≥7.0% to ≤11.0%
* Adult men or adult non-pregnant, non-breastfeeding women
* Body Mass Index (BMI) of ≥19.0 to ≤35.0 kilograms/square meter (kg/m^2)
* Stable weight (±5%) ≥3 months prior to screening

Exclusion Criteria:

* Have type 1 diabetes mellitus
* Have previous treatment with a glucagon-like peptide-1 (GLP-1) receptor agonist, GLP-1 analog, or any other incretin mimetic
* Have treatment with dipeptidyl peptidase-IV (DPP-IV) inhibitor, an alpha-glucosidase inhibitor (AGI), thiazolidinedione (TZD), or glinide
* Have gastric emptying abnormality
* Have cardiac disorder defined as unstable angina, myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention, heart failure, arrhythmia, transient ischemic attack, or stroke
* Have poorly controlled hypertension (systolic blood pressure above 160 millimeter of mercury[mmHg] or diastolic blood pressure above 95 mmHg)
* Have impaired liver function
* Have impaired kidney function
* Have history of chronic pancreatitis or acute pancreatitis
* Have a serum calcitonin ≥20 picograms per milliliter (pg/mL)
* Have a personal or family history of medullary C-cell hyperplasia, focal hyperplasia, carcinoma, or multiple endocrine neoplasia type 2 (MEN 2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 774 (Actual)
Dates: Start 2012-07; Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (29):
- China (20):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chengdu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chongqing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dalian
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guiyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harbin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hefei
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanchang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanning
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shenyang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shijiazhuang
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Xi'an
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Yangzhou
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Zhenjiang
- Mexico (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chihuahua City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Russia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chelyabinsk
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saint Petersburg
- South Korea (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucheon-si
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kyunggi-Do
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seoul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wŏnju

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Cai TT, Li HQ, Jiang LL, Wang HY, Luo MH, Su XF, Ma JH. Effects of GLP-1 Receptor Agonists on Bone Mineral Density in Patients with Type 2 Diabetes Mellitus: A 52-Week Clinical Study. Biomed Res Int. 2021 Sep 17;2021:3361309. doi: 10.1155/2021/3361309. eCollection 2021. PMID 34580638
- [Derived] Zhou Y, Zhu J, Wu H, Deng Y, Ji Q. Pancreatic Safety of Once-Weekly Dulaglutide in Chinese Patients with Type 2 Diabetes Mellitus: Subgroup Analysis by Potential Influencing Factors. Diabetes Ther. 2021 Oct;12(10):2677-2690. doi: 10.1007/s13300-021-01139-2. Epub 2021 Aug 28. PMID 34453682
- [Derived] Ma J, Zhang B, Hou J, Peng Y. Efficacy and Safety of Once Weekly Dulaglutide in East Asian Patients with Type 2 Diabetes: Subgroup Analysis by Potential Influential Factors. Diabetes Ther. 2021 Jan;12(1):211-222. doi: 10.1007/s13300-020-00955-2. Epub 2020 Nov 8. PMID 33161492
- [Derived] Kuang J, Zhu J, Liu S, Li Q. Efficacy and Safety of Once-Weekly Dulaglutide in Elderly Chinese Patients with Type 2 Diabetes: A Post Hoc Analysis of AWARD-CHN Studies. Diabetes Ther. 2020 Oct;11(10):2329-2339. doi: 10.1007/s13300-020-00910-1. Epub 2020 Aug 28. PMID 32857293
- [Derived] Guo L, Zhang B, Hou J, Zhou Z. Evaluation of Characteristics of Gastrointestinal Adverse Events with Once-Weekly Dulaglutide Treatment in Chinese Patients with Type 2 Diabetes: A Post Hoc Pooled Analysis of Two Randomized Trials. Diabetes Ther. 2020 Aug;11(8):1821-1833. doi: 10.1007/s13300-020-00869-z. Epub 2020 Jul 4. PMID 32621083
- [Derived] Yu M, Yuan GY, Zhang B, Wu HY, Lv XF. Efficacy and Safety of Dulaglutide by Baseline HbA1c in Chinese Patients with Type 2 Diabetes: A Post Hoc Analysis. Diabetes Ther. 2020 May;11(5):1147-1159. doi: 10.1007/s13300-020-00804-2. Epub 2020 Apr 10. PMID 32277401
- [Derived] Wang J, Li HQ, Xu XH, Kong XC, Sun R, Jing T, Ye L, Su XF, Ma JH. The Effects of Once-Weekly Dulaglutide and Insulin Glargine on Glucose Fluctuation in Poorly Oral-Antidiabetic Controlled Patients with Type 2 Diabetes Mellitus. Biomed Res Int. 2019 Dec 24;2019:2682657. doi: 10.1155/2019/2682657. eCollection 2019. PMID 31950036
- [Derived] Li Y, Li L, De Peng Y, Song GY, Ye SD, Du LY, Hou JN, Ji QH. Efficacy and Safety of Dulaglutide Versus Insulin Glargine in Chinese T2DM Patients: A Subgroup Analysis of a Randomized Trial (AWARD-CHN2). Diabetes Ther. 2019 Aug;10(4):1435-1452. doi: 10.1007/s13300-019-0646-y. Epub 2019 Jun 21. PMID 31228090

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a parallel-arm, non-inferiority study. Study treatment continued for up to 52 weeks and participants were randomized in a 1:1:1 ratio to one of the 3 treatment arms: 1.5 milligrams (mg) dulaglutide once-weekly , 0.75 mg dulaglutide once-weekly, or insulin glargine once-daily.
Groups:
- 1.5 mg Dulaglutide: 1.5 mg dulaglutide administered as 1 subcutaneous (SC) injection once-weekly added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea.
- 0.75 mg Dulaglutide: 0.75 mg dulaglutide administered as 1 SC injection once-weekly added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea.
- Insulin Glargine: Insulin glargine administered per dosing titration schedule as once daily SC injection at bedtime added to participant's pre-study prescribed dose of metformin and /or a sulfonylurea.
Period: Overall Study
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Started | 258 | 257 | 259
Received at Least One Dose of Study Drug | 258 | 257 | 259
Modified Intent-to-Treat Population | 253 | 252 | 250
Completed | 226 | 219 | 227
Not Completed | 32 | 38 | 32
Not completed — Adverse Event | 6 | 11 | 2
Not completed — Lost to Follow-up | 9 | 6 | 8
Not completed — Protocol Violation | 1 | 2 | 1
Not completed — Withdrawal by Subject | 15 | 17 | 17
Not completed — Physician Decision | 0 | 1 | 3
Not completed — Death | 1 | 0 | 0
Not completed — Sponsor Decision | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported for the modified intent-to-treat (mITT) population, who are all randomized participants with a baseline glycosylated hemoglobin (HbA1c) measurement, at least 1 post-baseline HbA1c measurement, and received at least 1 dose of study drug.
Groups:
- 1.5 mg Dulaglutide: 1.5 mg dulaglutide administered as 1 SC injection once-weekly added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea.
- Insulin Glargine: Insulin glargine administered per dosing titration schedule as once daily SC injection at bedtime added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea.
- Total: Total of all reporting groups
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine | Total
Number analyzed (Participants) | 253 | 252 | 250 | 755
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.03 (9.572) | 54.54 (10.006) | 55.44 (9.197) | 55.00 (9.593)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 109 | 111 | 338
  Male | 135 | 143 | 139 | 417
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14 | 14 | 13 | 41
  Asian | 213 | 209 | 209 | 631
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 26 | 29 | 28 | 83
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 200 | 196 | 195 | 591
  Korea, Republic of | 13 | 13 | 14 | 40
  Mexico | 22 | 24 | 24 | 70
  Russian Federation | 18 | 19 | 17 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at 26 Weeks
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. Least square (LS) means of change from baseline in HbA1c were calculated using a mixed-effects model for repeated measures (MMRM) with the change in HbA1c as the dependent variable and treatment, baseline HbA1c, country, oral antihyperglycemic medication (OAM) , visit, and treatment-by-visit interaction as fixed effects, and participant was the random effect.
Time Frame: Baseline, 26 Weeks
Population: Participants who were randomized, received at least one dose of study drug, and had evaluable HbA1c data at both baseline and post-baseline.
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 253 | 252 | 250
percentage of HbA1c | -1.73 (0.067) | -1.33 (0.067) | -1.16 (0.067)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — Analyses were based on a pre-defined non-inferiority margin of 0.4%; Mean Difference (Net) = -0.57, 95% CI 2-sided [-0.74 to -0.40]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — Analyses were based on a pre-defined non-inferiority margin of 0.4%; Mean Difference (Net) = -0.18, 95% CI 2-sided [-0.35 to -0.01]

2. Secondary Outcome: Change From Baseline in HbA1c at 52 Weeks
Description: HbA1c is a form of hemoglobin that is measured primarily to identify the average plasma glucose concentration over prolonged periods of time. LS means of change from baseline in HbA1c were calculated using a MMRM with the change in HbA1c as the dependent variable and treatment, baseline HbA1c, country, OAM, visit, and treatment-by-visit interaction as fixed effects, and participant was as the random effect.
Time Frame: Baseline, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of HbA1c
Groups:
- 1.5 mg Dulaglutide: 1.5 mg dulaglutide administered as one SC injection once-weekly added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea.
- 0.75 mg Dulaglutide: 0.75 mg dulaglutide administered as one SC injection once-weekly added to participant's pre-study prescribed dose of metformin and/or a sulfonylurea.
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 253 | 252 | 250
percentage of HbA1c | -1.47 (0.076) | -1.03 (0.076) | -0.89 (0.075)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — Analyses were based on a pre-defined non-inferiority margin of 0.4%; Mean Difference (Net) = -0.57, 95% CI 2-sided [-0.77 to -0.38]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Test type: Non-Inferiority or Equivalence — Analyses were based on a pre-defined non-inferiority margin of 0.4%; Mean Difference (Net) = -0.13, 95% CI 2-sided [-0.33 to -0.06]

3. Secondary Outcome: Percentage of Participants Attaining HbA1c of <7% or ≤6.5% at 26 Weeks and 52 Weeks
Description: The percentage of participants was calculated by dividing the number of participants reaching target HbA1c by the total number of participants analyzed, multiplied by 100.
Time Frame: Up to 26 and 52 weeks
Population: Participants who were randomized, received at least one dose of study drug, and had evaluable HbA1c data at both baseline and post-baseline. Missing endpoints were imputed with the last observation carried forward (LOCF) method.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 253 | 252 | 250
percentage of participants
  HbA1c <7%, Week 26 | 64.8 | 52.8 | 40.0
  HbA1c ≤6.5%, Week 26 | 51.4 | 38.9 | 21.6
  HbA1c <7%, Week 52 | 51.8 | 45.6 | 32.0
  HbA1c ≤6.5%, Week 52 | 37.2 | 31.3 | 17.2
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; <7.0% Week 26; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; <7.0 Week 26; Test type: Superiority or Other; p = 0.004, Fisher Exact
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; <=6.5% Week 26; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; <=6.5% Week 26; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 5: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; <7.0% Week 52; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 6: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; <7.0% Week 52; Test type: Superiority or Other; p = 0.002, Fisher Exact
Statistical Analysis 7: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; <=6.5% Week 52; Test type: Superiority or Other; p < 0.001, Fisher Exact
Statistical Analysis 8: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; <=6.5% Week 52; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: Change From Baseline in Fasting Blood Glucose (FBG) at 26 Weeks and 52 Weeks
Description: LS means of change from baseline were calculated using MMRM with the change in FBG as the dependent variable and treatment, baseline value, country, OAM, visit, and treatment-by-visit interaction as fixed effects, and participant was the random effect.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: millimoles per liter (mmol/L)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 253 | 252 | 250
millimoles per liter (mmol/L)
  Change from baseline in FBG, 26 Weeks | -2.35 (0.162) | -1.71 (0.161) | -2.59 (0.161)
  Change from baseline in FBG, 52 Weeks | -2.23 (0.166) | -1.53 (0.165) | -2.35 (0.164)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Week 26; Test type: Superiority or Other; p = 0.177, Mixed Models Analysis; Mean Difference (Net) = 0.24, 95% CI 2-sided [-0.11 to 0.59]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.88, 95% CI 2-sided [0.53 to 1.23]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Week 52; Test type: Superiority or Other; p = 0.518, Mixed Models Analysis; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.25 to 0.50]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.82, 95% CI 2-sided [0.45 to 1.20]

5. Secondary Outcome: Change From Baseline in 7-point Self-monitored Blood Glucose (SMBG) Profiles at 26 Weeks and 52 Weeks
Description: Participants were required to perform 7-point SMBG profiles on 2 separate, nonconsecutive days during the 2 weeks before randomization and Weeks 8, 14, 20, 26, 39, and 52 (or the Early Discontinuation Visit). SMBG measurements were taken using a plasma-equivalent blood glucose (BG) meter at 7 time points: morning pre-meal, morning 2 hours post-meal, mid-day pre-meal, mid-day 2 hours post-meal, evening pre-meal, evening 2 hours post-meal, and at bedtime. Mean and Week 26 and Week 52 was assessed in all treatment groups. LS means of change from baseline were calculated using MMRM with the change in 7-point SMBG as the dependent variable and treatment, baseline value, country, OAM, visit, and treatment-by-visit interaction as fixed effects, and participant was the random effect.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
mmol/L
  Morning pre-meal, Week 26 | -2.18 (0.104) | -1.89 (0.103) | -2.83 (0.103)
  Morning 2 hours post-meal, Week 26 | -3.81 (0.190) | -3.43 (0.188) | -3.32 (0.188)
  Mid-day pre-meal, Week 26 | -2.45 (0.159) | -2.07 (0.157) | -2.10 (0.157)
  Mid-day 2 hours post-meal, Week 26 | -3.16 (0.182) | -2.71 (0.179) | -2.11 (0.179)
  Evening pre-meal, Week 26 | -2.25 (0.150) | -1.74 (0.147) | -1.62 (0.148)
  Evening 2 hours post-meal, Week 26 | -3.00 (0.180) | -2.58 (0.178) | -2.11 (0.178)
  Bed time, Week 26 | -2.95 (0.170) | -2.51 (0.167) | -2.16 (0.167)
  Morning pre-meal, Week 52 | -2.06 (0.108) | -1.76 (0.108) | -2.83 (0.107)
  Morning 2 hours post-meal, Week 52 | -3.58 (0.201) | -3.25 (0.200) | -3.05 (0.197)
  Mid-day pre-meal, Week 52 | -2.37 (0.162) | -1.89 (0.162) | -1.94 (0.160)
  Mid-day 2 hours post-meal, Week 52 | -2.75 (0.187) | -2.61 (0.186) | -2.12 (0.184)
  Evening pre-meal, Week 52 | -2.15 (0.159) | -1.61 (0.158) | -1.51 (0.156)
  Evening 2 hours post-meal, Week 52 | -2.93 (0.183) | -2.54 (0.182) | -2.10 (0.180)
  Bed time, Week 52 | -2.90 (0.172) | -2.50 (0.171) | -1.91 (0.168)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Morning pre-meal, Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.65, 95% CI 2-sided [0.42 to 0.88]
Statistical Analysis 2: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Morning pre-meal, Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.94, 95% CI 2-sided [0.71 to 1.17]
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Morning 2-hours post-meal, Week 26; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.92 to -0.07]
Statistical Analysis 4: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Morning 2-hours post-meal, Week 26; Test type: Superiority or Other; p = 0.617, Mixed Models Analysis; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.53 to 0.32]
Statistical Analysis 5: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Mid-day pre-meal, Week 26; Test type: Superiority or Other; p = 0.055, Mixed Models Analysis; Mean Difference (Net) = -0.35, 95% CI 2-sided [-0.70 to 0.01]
Statistical Analysis 6: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Mid-day pre-meal, Week 26; Test type: Superiority or Other; p = 0.855, Mixed Models Analysis; Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.32 to 0.39]
Statistical Analysis 7: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Mid-day 2-hours post-meal, Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -1.05, 95% CI 2-sided [-1.46 to -0.64]
Statistical Analysis 8: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Mid-day 2-hours post-meal, Week 26; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Net) = -0.60, 95% CI 2-sided [-1.01 to -0.19]
Statistical Analysis 9: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Evening pre-meal, Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.63, 95% CI 2-sided [-0.97 to -0.29]
Statistical Analysis 10: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Evening pre-meal, Week 26; Test type: Superiority or Other; p = 0.489, Mixed Models Analysis; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.45 to 0.22]
Statistical Analysis 11: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Evening 2-hours post-meal, Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.89, 95% CI 2-sided [-1.30 to -0.48]
Statistical Analysis 12: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Evening 2-hours post-meal, Week 26; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis; Mean Difference (Net) = -0.47, 95% CI 2-sided [-0.88 to -0.06]
Statistical Analysis 13: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Bedtime, Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.79, 95% CI 2-sided [-1.17 to -0.41]
Statistical Analysis 14: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Bedtime, Week 26; Test type: Superiority or Other; p = 0.067, Mixed Models Analysis; Mean Difference (Net) = -0.35, 95% CI 2-sided [-0.73 to -0.03]
Statistical Analysis 15: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Morning pre-meal, Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.77, 95% CI 2-sided [0.52 to 1.01]
Statistical Analysis 16: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Morning pre-meal, Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 1.06, 95% CI 2-sided [0.82 to 1.31]
Statistical Analysis 17: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Morning 2-hours post-meal, Week 52; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; Mean Difference (Net) = -0.53, 95% CI 2-sided [-1.00 to -0.07]
Statistical Analysis 18: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Morning 2-hours post-meal, Week 52; Test type: Superiority or Other; p = 0.384, Mixed Models Analysis; Mean Difference (Net) = -0.21, 95% CI 2-sided [-0.67 to 0.26]
Statistical Analysis 19: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Mid-day pre-meal, Week 52; Test type: Superiority or Other; p = 0.024, Mixed Models Analysis; Mean Difference (Net) = -0.43, 95% CI 2-sided [-0.80 to -0.06]
Statistical Analysis 20: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Mid-day pre-meal, Week 52; Test type: Superiority or Other; p = 0.783, Mixed Models Analysis; Mean Difference (Net) = -0.05, 95% CI 2-sided [-0.32 to 0.42]
Statistical Analysis 21: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Mid-day 2-hours post-meal, Week 52; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Net) = -0.63, 95% CI 2-sided [-1.07 to -0.20]
Statistical Analysis 22: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Mid-day 2-hours post-meal, Week 52; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; Mean Difference (Net) = -0.48, 95% CI 2-sided [-0.92 to -0.05]
Statistical Analysis 23: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Evening pre-meal, Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.64, 95% CI 2-sided [-1.01 to -0.27]
Statistical Analysis 24: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Evening pre-meal, Week 52; Test type: Superiority or Other; p = 0.603, Mixed Models Analysis; Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.47 to 0.27]
Statistical Analysis 25: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Evening 2-hours post-meal, Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.83, 95% CI 2-sided [-1.26 to -0.41]
Statistical Analysis 26: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Evening 2-hours post-meal, Week 52; Test type: Superiority or Other; p = 0.039, Mixed Models Analysis; Mean Difference (Net) = -0.45, 95% CI 2-sided [-0.87 to -0.02]
Statistical Analysis 27: Comparison: 1.5 mg Dulaglutide vs Insulin Glargine; Bedtime, Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.99, 95% CI 2-sided [-1.39 to -0.60]
Statistical Analysis 28: Comparison: 0.75 mg Dulaglutide vs Insulin Glargine; Bedtime, Week 52; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mean Difference (Net) = -0.59, 95% CI 2-sided [-0.98 to -0.20]

6. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment 2 Steady-state Beta (β)- Cell Function (HOMA2-%B) at 26 Weeks and 52 Weeks
Description: The updated Homeostasis Model Assessment (HOMA2) was used to quantify steady state beta-cell function (%B). HOMA2-%B is a computer model that uses fasting plasma insulin and glucose concentrations to estimate %B as a percentage of a normal reference population. LS means were calculated using a homeostasis model assessment with change from baseline in HOMA-%B as a covariate and country, baseline measurement, OAM, and treatment as fixed effects.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: Participants who were randomized, received at least one dose of study drug, and had evaluable HbA1c data at both baseline and post-baseline. Missing endpoints were imputed with the LOCF method. HOMA2 was not evaluated for insulin glargine, as the use of this model has not been validated in participants treated with insulin.
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2-%B
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 253 | 252
percentage of HOMA2-%B
  Insulin-Based HOMA2-%B, 26 Weeks | 34.41 (3.831) | 31.17 (3.761)
  Insulin-Based HOMA2-%B, 52 Weeks | 45.12 (4.147) | 36.64 (4.061)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%B, Dula 1.5 mg, Week 26; Test type: Superiority or Other; p = 0.352, Mixed Models Analysis; Mean Difference (Net) = 34.41, Standard Error of Mean 3.831
Statistical Analysis 2: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%B, Dula 0.75 mg, Week 26; Test type: Superiority or Other; p = 0.352, Mixed Models Analysis; Mean Difference (Net) = 31.17, Standard Error of Mean 3.761
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%B, Dula 1.5, Week 52; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; Mean Difference (Net) = 45.12, Standard Error of Mean 4.147
Statistical Analysis 4: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%B, Dula 0.75 mg, Week 52; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; Mean Difference (Net) = 36.64, Standard Error of Mean 4.061

7. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment 2 Insulin Sensitivity - Cell Function (HOMA2-%S) at 26 Weeks and 52 Weeks
Description: The HOMA2 was used to estimate the steady-state insulin sensitivity (%S). HOMA2-S is a computer model that uses fasting plasma insulin and glucose concentrations to estimate insulin sensitivity (%S) as a percentage of the normal reference population. LS means were calculated using an homeostasis model assessment with change from baseline in HOMA-%S as a covariate and country, baseline measurement, OAM, and treatment as fixed effects.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: percentage of HOMA2-%S
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide
Number analyzed (Participants) | 253 | 252
percentage of HOMA2-%S
  Insulin-Based HOMA2-%S, Week 26 | -6.86 (3.649) | -10.03 (3.591)
  Insulin-Based HOMA2-%S, Week 52 | -10.19 (3.677) | -12.32 (3.609)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%S, Dula 1.5 mg, Week 26; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; Mean Difference (Net) = 36.57, Standard Error of Mean 2.977
Statistical Analysis 2: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%S, Dula 0.75 mg, Week 26; Test type: Superiority or Other; p = 0.025, Mixed Models Analysis; Mean Difference (Net) = 30.42, Standard Error of Mean 2.940
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%S, Dula 1.5 mg, Week 52; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; Mean Difference (Net) = 41.02, Standard Error of Mean 2.900
Statistical Analysis 4: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; HOMA2-%S, Dula 0.75 mg, Week 52; Test type: Superiority or Other; p = 0.029, Mixed Models Analysis; Mean Difference (Net) = 35.19, Standard Error of Mean 2.864

8. Secondary Outcome: Rate of Hypoglycemic Events
Description: Hypoglycemic events (HE) were classified as documented symptomatic hypoglycemia, asymptomatic hypoglycemia, severe hypoglycemia, and probable symptomatic hypoglycemia. The 1-year adjusted rate of HEs was summarized cumulatively at 26 weeks and 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 weeks and 52 weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: events per participant per year
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
events per participant per year
  1-year Rate of HE, Week 26 | 1.27 (4.485) | 0.98 (4.202) | 2.13 (6.724)
  Severe HE Week 26 | NA (NA) — Data not available because no severe hypoglycemic episodes occurred. | NA (NA) — Data not available because no severe hypoglycemic episodes occurred. | NA (NA) — Data not available because no severe hypoglycemic episodes occurred.
  Nocturnal HE Week 26 | 0.19 (0.904) | 0.13 (0.762) | 0.38 (1.444)
  1-year Rate of HE, Week 52 | 0.89 (3.777) | 0.80 (3.914) | 1.92 (6.983)
  Severe HE Week 52 | NA (NA) — Data not available because no severe hypoglycemic episodes occurred. | NA (NA) — Data not available because no severe hypoglycemic episodes occurred. | NA (NA) — Data not available because no severe hypoglycemic episodes occurred.
  Nocturnal HE Week 52 | 0.11 (0.488) | 0.10 (0.551) | 0.31 (1.261)

9. Secondary Outcome: Number of Self-reported Hypoglycemic Events
Description: Hypoglycemic events (HE) were classified as severe (defined as episodes requiring the assistance of another person to actively administer resuscitative actions), documented symptomatic (defined as any time a participant felt that he/she was experiencing symptoms and/or signs associated with hypoglycemia, and had a plasma glucose level of less than or equal to 3.9 millimoles/liter [mmol/L]), asymptomatic (defined as events not accompanied by typical symptoms of hypoglycemia but with a measured plasma glucose of less than or equal to 3.9 mmol/L), nocturnal (defined as any hypoglycemic event that occurred between bedtime and waking), or probable symptomatic (defined as events during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination). The number of self-reported hypoglycemic events was summarized cumulatively at 52 weeks. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 26 Weeks and 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
percentage of participants
  Total HE Week 26 | 19.4 | 16.7 | 29.6
  Severe HE Week 26 | 0.0 | 0.0 | 0.0
  Nocturnal HE Week 26 | 6.2 | 3.9 | 11.1
  Documented Symptomatic Week 26 | 11.2 | 7.8 | 17.0
  Asymptomatic HE Week 26 | 10.1 | 8.2 | 14.2
  Probable HE Week 26 | 4.3 | 5.1 | 7.5
  Total HE Week 52 | 22.5 | 19.8 | 34.8
  Severe HE Week 52 | 0.0 | 0.0 | 0.0
  Nocturnal HE Week 52 | 7.0 | 4.3 | 13.8
  Documented Symptomatic HE Week 52 | 12.4 | 9.7 | 20.6
  Asymptomatic HE Week 52 | 12.0 | 10.1 | 19.4
  Probable HE Week 52 | 4.7 | 5.4 | 8.3

10. Secondary Outcome: Change From Baseline to 26 Weeks and 52 Weeks on Blood Pressure (BP)
Description: Seated systolic blood pressure (SBP) and seated diastolic blood pressure (DBP) were measured. LS means of change from baseline were calculated using a MMRM with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: millimeters of mercury (mmHg)]
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
millimeters of mercury (mmHg)]
  SBP 26 Weeks | -5.53 (12.037) | -2.77 (11.920) | -2.22 (12.743)
  DBP 26 Weeks | -1.58 (7.842) | -0.92 (7.898) | -1.61 (8.417)
  SBP 52 Weeks | -2.18 (11.134) | -0.61 (12.081) | -0.25 (11.717)
  DBP 52 Weeks | -0.19 (7.542) | 0.44 (7.582) | -1.13 (8.810)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 26 SBP; Test type: Superiority or Other; p = 0.008, Mixed Models Analysis — Overall p-value
Statistical Analysis 2: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 26 DBP; Test type: Superiority or Other; p = 0.584, Mixed Models Analysis — Overall p-value
Statistical Analysis 3: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 52 SBP; Test type: Superiority or Other; p = 0.169, Mixed Models Analysis — Overall p-value
Statistical Analysis 4: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 52 DBP; Test type: Superiority or Other; p = 0.110, Mixed Models Analysis — Overall p-value

11. Secondary Outcome: Change From Baseline at 26 Weeks and 52 Weeks on Pulse Rate
Description: Seated pulse rate was measured. LS means of change from baseline were calculated using a MMRM with treatment, country, visit, and treatment-by-visit interaction as fixed effects and baseline as a covariate.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: beats per minute (bpm)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
beats per minute (bpm)
  Change From Baseline on Pulse rate at Week 26 | 4.63 (8.681) | 0.65 (8.631) | -0.86 (9.546)
  Change From Baseline on Pulse rate at Week 52 | 4.18 (8.336) | 3.18 (8.917) | 0.07 (8.205)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Overall p-value
Statistical Analysis 2: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Overall p-value

12. Secondary Outcome: Change From Baseline in Electrocardiogram Parameters, Fridericia Corrected QT (QTcF) Interval and PR Interval
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave and was calculated from electrocardiogram (ECG) data using Fridericia's formula: QTc = QT/RR^0.33. Corrected QT (QTc) is the QT interval corrected for heart rate and RR, which is the interval between two R waves. PR is the interval between the P wave and the QRS complex.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: millisecond (msec)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
millisecond (msec)
  QTcF Interval 26 Weeks | -1.65 (13.157) | 0.76 (11.643) | 2.56 (11.911)
  PR Interval 26 Weeks | 3.09 (1.700) | 2.88 (10.801) | -0.86 (10.272)
  QTcF Interval 52 Weeks | 0.55 (11.209) | 1.19 (12.165) | 4.03 (11.446)
  PR Interval 52 Weeks | 3.60 (12.425) | 3.55 (11.526) | 0.63 (11.861)

13. Secondary Outcome: Change From Baseline in Electrocardiogram Parameters, Heart Rate (HR)
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
beats per minute (bpm)
  Week 26 | 6.13 (8.924) | 3.77 (9.002) | -0.46 (9.329)
  Week 52 | 5.04 (8.223) | 3.40 (7.986) | 0.43 (8.060)

14. Secondary Outcome: Change From Baseline in Pancreatic Enzymes
Description: Amylase (total and pancreas-derived) and lipase concentrations were measured
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug. Last observation carried forward (LOCF) was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: Units/Liter (U/L)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
Units/Liter (U/L)
  Amylase, Total 26 Weeks | 7.50 (18.755) | 7.54 (22.388) | -0.37 (18.196)
  Amylase, pancreas derived 26 Weeks | 5.83 (14.607) | 5.14 (19.360) | -0.21 (11.287)
  Lipase 26 Weeks | 11.00 (34.134) | 10.67 (39.989) | -2.74 (21.818)
  Amylase, Total 52 Weeks | 7.82 (16.250) | 6.42 (20.675) | 0.64 (18.696)
  Amylase, pancreas derived 52 Weeks | 5.48 (12.449) | 4.05 (15.490) | -0.49 (12.576)
  Lipase 52 Weeks | 10.76 (27.360) | 9.64 (33.715) | -3.66 (20.484)

15. Secondary Outcome: Change From Baseline in Serum Calcitonin
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug. Only pre-rescue measurements were used. LOCF was used to impute missing postbaseline values. If there were no data after the date of randomization, the endpoint was considered missing.
Measure: Mean (Standard Deviation); unit: picomole/liter
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
picomole/liter
  Week 26 | 0.01 (0.240) | -0.07 (0.289) | 0.02 (0.256)
  Week 52 | -0.03 (0.279) | -0.08 (0.325) | -0.05 (0.306)

16. Secondary Outcome: Number of Participants With Adjudicated Cardiovascular (CV) Events
Description: Deaths and nonfatal cardiovascular adverse events were adjudicated by a committee of physicians with cardiology expertise external to the Sponsor. The nonfatal cardiovascular events subjected to adjudication included myocardial infarction, hospitalization for unstable angina, hospitalization for heart failure, coronary interventions (such as coronary artery bypass graft or percutaneous coronary intervention), and cerebrovascular events including cerebrovascular accident (stroke) and transient ischemic attack. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Number; unit: participants with adjudicated CV events
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
participants with adjudicated CV events | 6 | 2 | 2

17. Secondary Outcome: Number of Participants With Adjudicated Pancreatitis
Description: The number of participants with pancreatitis confirmed by adjudication is summarized. Events of pancreatitis (including suspected pancreatitis and severe or serious abdominal pain) were adjudicated by a committee of expert physicians external to the Sponsor. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
participants | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in Body Weight
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: kilogram (kg)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
kilogram (kg)
  Week 26 | -1.47 (0.197) | -0.88 (0.197) | 0.97 (0.198)
  Week 52 | -1.08 (0.201) | -0.76 (0.202) | 1.35 (0.201)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — Week 26
Statistical Analysis 2: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

19. Secondary Outcome: Change in Body Mass Index
Description: Body mass index is an estimate of body fat based on body weight divided by height squared.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: kilogram/square meter (kg/m2)
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
kilogram/square meter (kg/m2)
  Week 26 | -0.53 (0.071) | -0.32 (0.071) | 0.37 (0.071)
  Week 52 | -0.40 (0.072) | -0.27 (0.072) | 0.52 (0.072)
Statistical Analysis 1: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide; Week 26; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis
Statistical Analysis 2: Comparison: 1.5 mg Dulaglutide vs 0.75 mg Dulaglutide vs Insulin Glargine; Week 52; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis

20. Secondary Outcome: Percentages of Participants Developing Treatment-Emergent Dulaglutide Anti-drug Antibody (ADA)
Description: Number of participants with treatment emergent (TE) dulaglutide anti-drug antibodies from postbaseline to follow up were summarized. A participant was considered to have TE dulaglutide ADA if the participant had at least one titer that was treatment-emergent relative to baseline, defined as a 4-fold or greater increase in titer from baseline measurement.
Time Frame: Baseline through 52 Weeks
Population: Participants in the safety population who were randomized and received at least one dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
Percentage of participants
  Participants with >=1 TE Dula ADA | 3.9 | 4.3 | 1.6
  Participants with TE Dula ADA and Neutralizing | 0.8 | 1.6 | 0.0

21. Secondary Outcome: EQ-5D Health State Score Responses
Description: The EQ-5D questionnaire is a widely used, generic questionnaire that assesses health-related quality of life. It consists of 2 parts. The first part assesses 5 dimensions associated with quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 3 possible levels of response: no problem, some problem, and extreme problem. Additional categories of response include ambiguous and missing. The number of participants per each of the 3 response categories is summarized for each of the 5 dimensions.
Time Frame: Baseline, 26 Weeks, 52 Weeks
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
participants
  Mobility - no problem Week 26 | 219 | 215 | 210
  Mobility - some problem Week 26 | 7 | 16 | 20
  Mobility - extreme problem Week 26 | 0 | 0 | 0
  Mobility - missing Week 26 | 4 | 1 | 4
  Self-care - no problem Week 26 | 223 | 227 | 224
  Self-care - some problem Week 26 | 0 | 0 | 0
  Self-care - extreme problem Week 26 | 0 | 0 | 0
  Self-care - missing Week 26 | 4 | 1 | 4
  Usual activities - no problems Week 26 | 219 | 220 | 218
  Usual activities - some problems Week 26 | 7 | 11 | 11
  Usual activities - extreme problems Week 26 | 0 | 0 | 0
  Usual activities - missing Week 26 | 4 | 1 | 4
  Pain/Discomfort - no problems Week 26 | 193 | 201 | 188
  Pain/Discomfort - some problems Week 26 | 32 | 30 | 37
  Pain/Discomfort - ambiguous | 0 | 0 | 0
  Pain/Discomfort - missing Week 26 | 4 | 1 | 4
  Anxiety/Depression - no problems Week 26 | 208 | 204 | 203
  Anxiety/Depression - some problems Week 26 | 19 | 27 | 26
  Anxiety/Depression - extreme problems Week 26 | 0 | 0 | 1
  Anxiety/Depression - missing Week 26 | 4 | 1 | 4
  Mobility - no problems Week 52 | 218 | 207 | 214
  Mobility - some problems Week 52 | 8 | 14 | 16
  Mobility - extreme problems Week 52 | 0 | 1 | 0
  Mobility - missing Week 52 | 0 | 0 | 1
  Self-care - no problems Week 52 | 224 | 215 | 223
  Self-care - some problems Week 52 | 2 | 7 | 7
  Self-care - extreme problems Week 52 | 0 | 0 | 0
  Self-care - missing Week 52 | 0 | 0 | 1
  Usual Activities - no problems Week 52 | 219 | 211 | 219
  Usual Activities - some problems Week 52 | 6 | 10 | 11
  Usual Activities - extreme problems Week 52 | 1 | 1 | 0
  Usual Activities - missing Week 52 | 0 | 0 | 1
  Pain/Discomfort - no problems Week 52 | 191 | 188 | 185
  Pain/Discomfort - some problems Week 52 | 34 | 33 | 43
  Pain/Discomfort - extreme problems Week 52 | 1 | 1 | 1
  Pain/Discomfort - missing Week 52 | 0 | 0 | 1
  Anxiety/Depression - no problems Week 52 | 205 | 207 | 201
  Anxiety/Depression - some problems Week 52 | 21 | 15 | 29
  Anxiety/Depression - extreme problems Week 52 | 0 | 0 | 0
  Anxiety/Depression - missing Week 52 | 0 | 0 | 1

22. Secondary Outcome: Change From Baseline in EQ-5D Visual Analog Scale Score
Description: The EQ-5D is a generic, multidimensional, health-related, quality-of-life instrument. Overall health state score was self-reported using a visual analogue scale (VAS) marked on a scale of 0 to 100 with 0 representing worst imaginable health state and 100 representing best imaginable health state. LS means of change from baseline were calculated using ANCOVA and adjusted by treatment, country, and baseline.
Time Frame: Baseline, 26 weeks, 52 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Number analyzed (Participants) | 258 | 257 | 253
units on a scale
  Week 26 | 1.08 (12.644) | 1.67 (13.456) | 1.41 (10.885)
  Week 52 | 2.65 (12.029) | 2.34 (14.003) | 2.55 (12.257)

ADVERSE EVENTS:
Arm/Group | 1.5 mg Dulaglutide | 0.75 mg Dulaglutide | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 24/258 | 15/257 | 9/253
Other Adverse Events (participants affected / at risk) | 184/258 | 188/257 | 157/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=258) | 0.75 mg Dulaglutide (N=257) | Insulin Glargine (N=253)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gallbladder empyema (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (2) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pulmonary tuberculoma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Comminuted fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Gun shot wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/119 (0) | 1/113 (1) | 0/112 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhagic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Perinephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 1.5 mg Dulaglutide (N=258) | 0.75 mg Dulaglutide (N=257) | Insulin Glargine (N=253)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Microcytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 3 (3) | 2 (2) | 2 (2)
Extrasystoles (Cardiac disorders) | 1 (2) | 1 (1) | 0 (0)
Left ventricular hypertrophy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Thyroid mass (Endocrine disorders) | 3 (3) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinopathy (Eye disorders) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 4 (4) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 5 (6) | 3 (4) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 18 (29) | 13 (16) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (6) | 3 (4) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 1 (1) | 3 (5)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (11) | 8 (8) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 43 (92) | 28 (51) | 7 (7)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 5 (6) | 8 (11) | 2 (2)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Eructation (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 4 (5) | 1 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric dilatation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Gastric disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (3) | 4 (4)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (7) | 1 (1) | 1 (2)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Intestinal polyp (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 27 (47) | 14 (21) | 2 (2)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Regurgitation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 16 (23) | 6 (6) | 2 (2)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 3 (3) | 0 (0)
Chest pain (General disorders) | 1 (2) | 5 (5) | 0 (0)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0)
Discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (2) | 1 (1)
Hunger (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Induration (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 1 (19) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 2 (2)
Nodule (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 3 (5)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 4 (4)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0)
Cholecystitis chronic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 1 (1) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic fibrosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 4 (4) | 3 (3)
Hepatic steatosis (Hepatobiliary disorders) | 3 (3) | 3 (3) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Liver injury (Hepatobiliary disorders) | 1 (1) | 4 (4) | 1 (1)
Non-alcoholic fatty liver (Hepatobiliary disorders) | 3 (3) | 7 (7) | 2 (2)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Post cholecystectomy syndrome (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 2 (2) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) | 2 (2)
Immunodeficiency (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Asymptomatic bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Cat scratch disease (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Conjunctivitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 4 (5) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 3 (4) | 3 (3)
Laryngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 18 (22) | 17 (23) | 22 (29)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 5 (5)
Pharyngitis bacterial (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis chronic (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Tracheobronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (9) | 10 (11) | 13 (15)
Urinary tract infection (Infections and infestations) | 13 (15) | 14 (14) | 11 (11)
Vaginal infection (Infections and infestations) | 2/119 (3) | 0/113 (0) | 0/112 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Exposure via father (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Albumin urine present (Investigations) | 0 (0) | 0 (0) | 2 (2)
Amylase abnormal (Investigations) | 0 (0) | 1 (3) | 1 (1)
Amylase increased (Investigations) | 7 (10) | 5 (13) | 1 (1)
Bacterial test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood cholesterol increased (Investigations) | 6 (6) | 6 (6) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood potassium abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 2 (3)
Blood triglycerides (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 4 (4) | 6 (6) | 3 (4)
Blood uric acid increased (Investigations) | 1 (1) | 0 (0) | 3 (3)
Blood urine (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0) | 2 (2)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Calcium ionised increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Carbohydrate antigen 19-9 increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Creatinine renal clearance increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Crystal urine present (Investigations) | 2 (3) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram low voltage (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram t wave abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 4 (4) | 0 (0)
Glucose urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Glucose urine present (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart rate increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
High density lipoprotein decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase abnormal (Investigations) | 0 (0) | 1 (3) | 1 (1)
Lipase increased (Investigations) | 27 (35) | 18 (23) | 2 (2)
Low density lipoprotein increased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Pancreatic enzymes increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine (Investigations) | 1 (1) | 0 (0) | 0 (0)
Protein urine present (Investigations) | 0 (0) | 1 (1) | 2 (2)
Urine albumin/creatinine ratio increased (Investigations) | 2 (2) | 4 (4) | 4 (4)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 19 (22) | 14 (19) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Dyslipidaemia (Metabolism and nutrition disorders) | 9 (10) | 6 (6) | 9 (10)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 46 (49) | 50 (54) | 47 (48)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (7) | 4 (4)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypolipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (8) | 1 (2)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/119 (0) | 2/113 (2) | 2/112 (2)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic autonomic neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Diabetic neuropathy (Nervous system disorders) | 1 (1) | 2 (2) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 5 (6) | 3 (3)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 8 (9) | 8 (8) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 3 (4) | 1 (1) | 5 (6)
Lacunar infarction (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Poor quality sleep (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1)
Albuminuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Diabetic nephropathy (Renal and urinary disorders) | 1 (1) | 5 (5) | 5 (5)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 3 (3) | 2 (2)
Hypertensive nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperuricosuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Microalbuminuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 3 (3) | 0 (0)
Nephroptosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Renal cyst (Renal and urinary disorders) | 1 (1) | 3 (3) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1/139 (1) | 0/144 (0) | 0/141 (0)
Endometrial thickening (Reproductive system and breast disorders) | 0/119 (0) | 2/113 (2) | 0/112 (0)
Menstrual disorder (Reproductive system and breast disorders) | 1/119 (1) | 0/113 (0) | 0/112 (0)
Polycystic ovaries (Reproductive system and breast disorders) | 0/119 (0) | 1/113 (1) | 0/112 (0)
Prostatitis (Reproductive system and breast disorders) | 0/139 (0) | 1/144 (1) | 0/141 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 3 (3)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Urticaria contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal polypectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Lung lobectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Modified radical mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Retinal laser coagulation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic vascular disorder (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 20 (20) | 28 (28) | 19 (19)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days